CLINICAL TRIAL: NCT02637323
Title: An Open-label, Single Administration Study to Characterize the Systemic Pharmacokinetics and Local Extent and Duration of Exposure of Triamcinolone Acetonide From FX006 in Patients With Osteoarthritis of the Knee
Brief Title: Study to Characterize the PK and Local Extent and Duration of Exposure From FX006 in Patients With OA of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2015-009
Record Dates: First submitted 2015-12-07; First posted 2015-12-22 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; pain; corticosteroid; intra-articular; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FX006 32 mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 32 mg
- TCA IR 40 mg (Active Comparator): Commercially available triamcinolone acetonide, single 1 mL intra-articular (IA) injection Immediate-release formulation
  Interventions: Drug: TCA IR 40

INTERVENTIONS:
Drug: FX006 32 mg — Single 5 mL IA injection
  Other Names: Zilretta
  Arms: FX006 32 mg
Drug: TCA IR 40 — Single 1 mL IA injection
  Other Names: Kenalog®-40 Injection; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
The objectives of this study were to characterize the local extent and duration of exposure of TA from FX006 and TCA IR, characterize the systemic PK of FX006 and TCA IR, and assess the safety and general tolerability of a single 5 mL IA injection of 32 mg FX006 relative to 40 mg of TCA IR in patients with OA of the knee.

DETAILED DESCRIPTION:
This study employed an open-label, single administration design and was conducted in male and female patients ≥40 years of age with OA of the knee.

Patients were enrolled sequentially with at least 10 patients per cohort as follows:

Cohort A: FX006 32 mg, Final Visit at Week 20 Cohort B: FX006 32 mg, Final Visit at Week 16 Cohort C: FX006 32 mg, Final Visit at Week 12 Cohort D: FX006 32 mg, Final Visit at Week 6 Cohort E: FX006 32 mg, Final Visit at Week 1 Cohort F: TCA IR 40 mg, Final Visit Week 6

Each patient was screened to confirm eligibility and assigned to a cohort on Day 1/baseline. Each patient was evaluated for safety during his/her participation in the study at 6, 12, 16, or 20 weeks following a single IA injection depending on the assigned Cohort, and plasma and synovial fluid was collected for drug concentration measurements.

Safety and tolerability was assessed by physical examinations, index knee examinations, vital signs, clinical laboratory evaluations, and adverse events (AEs).

No efficacy assessments were employed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Symptoms associated with OA of the knee for ≥ 6 months prior to Screening (patient reported is acceptable)
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA
* Index knee pain for >15 days over the last month (as reported by the patient)
* Body mass index (BMI) ≤ 40 kg/m2
* Ambulatory and in good general health

Exclusion Criteria:

* Fibromyalgia, Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of infection in the index knee joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee within 1 month of Screening
* Presence of surgical hardware or other foreign body in the index knee
* Unstable joint within 12 months of Screening
* IA corticosteroid (investigational or marketed) in any joint within 6 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Intravenous or Intramuscular corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Any other IA investigational drug/biologic use within 6 months of Screening or 5 half-lives (whichever is longer)
* Prior use of FX006
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (4):
- United States (4):
  - Canoga Park, California
  - San Diego, California
  - Hialeah, Florida
  - Duncansville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for study eligibility at four (4) study centers in the United States (US).
Pre-assignment Details: Patients were enrolled sequentially with at least 10 patients per Cohort. Subjects were enrolled within 14 days of Screening.
Groups:
- FX006 32 mg: 63 subjects received FX006 32 mg as a single 5 mL IA injection
- TCA IR 40 mg: 18 subjects received TCA IR 40 mg as a single 1 mL IA injection
Period: Overall Study
Arm/Group | FX006 32 mg | TCA IR 40 mg
Started | 63 | 18
Completed | 61 | 17
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TCA IR 40 mg: Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 32 mg | TCA IR 40 mg | Total
Number analyzed (Participants) | 63 | 18 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (8.16) | 61.9 (7.68) | 61 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 13 | 45
  Male | 31 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Synovial Fluid Drug Concentrations (pg/mL) by Time Point Pooled Across FX006 Cohorts and TCA IR in Synovial Fluid
Description: All baseline (pre-treatment) values and all post-baseline values recorded as below LLOQ (<50 pg/mL) were set to zero. Geometric mean summary statistics were computed on adjusted concentration values. One (1) was added to each concentration value observed. BLQ values for the computation of geometric mean are included in the summary with a value of 1 (0+1).
Time Frame: Up to 20 Weeks
Population: All patients who received study drug and had synovial fluid obtained at the Synovial Fluid Visit and assayed for drug concentration levels.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 17 | 8
pg/mL
  Baseline (pre-treatment): number analyzed (Participants) | 17 | 5
  Baseline (pre-treatment) | 1.0 [1.00 to 1.00] | 1.0 [1.00 to 1.00]
  Week 1: number analyzed (Participants) | 8 | 0
  Week 1 | 231328.9 [56460.40 to 947798.36] |
  Week 6: number analyzed (Participants) | 6 | 8
  Week 6 | 3590.0 [32.89 to 391914.74] | 7.7 [0.31 to 191.34]
  Week 12: number analyzed (Participants) | 9 | 0
  Week 12 | 290.6 [15.67 to 5390.53] |
  Week 16: number analyzed (Participants) | 2 | 0
  Week 16 | 1.0 [1.00 to 1.00] |
  Week 20: number analyzed (Participants) | 4 | 0
  Week 20 | 1.0 [1.00 to 1.00] |

2. Secondary Outcome: Plasma Drug Concentrations (pg/mL) by Time Pooled Across FX006 Cohorts and TCA IR 40 mg Cohort
Description: All baseline (pre-treatment) values and all post-baseline values that are recorded as below LLOQ were set to zero for analysis and were included in the descriptive mean calculations. Values below LLOQ were not included in geometric mean calculations.
Time Frame: Up to 20 Weeks
Population: All patients who received study drug and had at least one post-baseline plasma sample obtained and assayed for drug concentration levels.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- FX006 32 mg: Single 5mL IA injection
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 60 | 18
pg/mL
  Day 1 - Hour 1 | 670.0 [558.42 to 803.97] | 6968.8 [3329.00 to 14588.36]
  Day 1 - Hour 2 | 736.5 [630.01 to 861.03] | 8494.7 [3954.18 to 18248.99]
  Day 1 - Hour 4 | 759.5 [641.69 to 898.87] | 9628.8 [4420.47 to 20973.81]
  Day 1 - Hour 6 | 747.1 [630.45 to 885.28] | 9314.3 [4423.76 to 19611.37]
  Day 1 - Hour 8 | 740.2 [625.13 to 876.36] | 8421.3 [4166.33 to 17021.86]
  Day 1 - Hour 10 | 720.7 [611.37 to 849.66] | 7439.3 [3845.19 to 14392.79]
  Day 1 - Hour 12 | 706.6 [600.15 to 831.91] | 6678.7 [3535.07 to 12617.78]
  Day 2 - Hour 24 | 836.4 [703.47 to 994.33] | 4991.1 [2851.47 to 8736.28]
  Week 1: number analyzed (Participants) | 11 | 0
  Week 1 | 600.9 [382.79 to 943.25] |
  Week 6: number analyzed (Participants) | 54 | 17
  Week 6 | 118.6 [99.93 to 140.87] | 149.4 [69.70 to 320.32]
  Week 12: number analyzed (Participants) | 15 | 0
  Week 12 | 53.7 [30.46 to 94.74] |
  Week 16: number analyzed (Participants) | 15 | 0
  Week 16 | 73.8 [28.74 to 189.31] |
  Week 20: number analyzed (Participants) | 8 | 0
  Week 20 | 108.2 [2.30 to 5090.25] |

3. Other Pre Specified Outcome: Plasma Pharmacokinetic Parameters for FX006 and TCA IR
Time Frame: Up to 20 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following IA administration on Baseline/Day 1 up to 20 weeks.
Groups:
- FX006 32 mg: Single 5 mL intra-articular injection
  FX006: Sustained Release Steroid
- TCA IR 40 mg: Commercially available triamcinolone acetonide, single 1 mL intra-articular injection
  TCA IR: Immediate Release Steroid
Arm/Group | FX006 32 mg | TCA IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/18
Other Adverse Events (participants affected / at risk) | 7/63 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=63) | TCA IR 40 mg (N=18)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=63) | TCA IR 40 mg (N=18)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Weight Increased (Investigations) | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Hypertension (Vascular disorders) | 2 (2) | 0
Flushing (Vascular disorders) | 0 | 2 (2)

LIMITATIONS AND CAVEATS:
Subsequent to completion of clinical studies extensive testing was performed to assess the actual FX006 dose delivered. It was determined that the FX006 delivered dose to the patient from an FX006 40 mg vial is 32 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes